CLINICAL TRIAL: NCT03726476
Title: Randomized Trial on Expectations and Pain Control Advancement In surgeRy: The REPAIR Trial
Brief Title: Expectations and Pain Control Advancement In surgeRy: The REPAIR Trial
Acronym: REPAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Peter C Jeppson, Principal Investigator, Assistant Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-262
Record Dates: First submitted 2018-07-13; First posted 2018-10-31 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-02

CONDITIONS: Abuses Over-The-Counter/Prescription Medications; Pain, Postoperative; Opioid Use; Physical Activity; Patient Dependence on
MeSH Terms: conditions — Pain, Postoperative; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Centered pre-op education (Experimental): Patient centered pre-operative education and patient centered post-operative care.
  Interventions: Behavioral: Patient centered pre-op education
- Routine Pre-op education (Active Comparator): Participants will receive routine pre-operative education and post-op will receive a standardized number of narcotics
  Interventions: Behavioral: routine preop education

INTERVENTIONS:
Behavioral: Patient centered pre-op education — To implement a patient centered education intervention to evaluate post-op narcotic use.
  Arms: Patient Centered pre-op education
Behavioral: routine preop education — To implement routine patient education intervention to evaluate post-op narcotic use.
  Arms: Routine Pre-op education

SUMMARY:
This is a randomized control trial that aims to evaluate whether patient-centered education, compared to routine education, decreases narcotic consumption without interfering with return to physical activity following hospital discharge. In addition, it will test whether patient-centered education decreases the quantity of narcotics prescribed and/or increases patient satisfaction and preparedness.

DETAILED DESCRIPTION:
Opioid use disorder is a national health emergency. Opioid prescribing practices to treat post-operative pain have contributed to the problem. This study seeks to explore the effects of changing pre-operative education & increasing patient input regarding post-operative receipt of opioids. The study will explore the effects that change in pre-operative education may have on post-operative opioid consumption juxtaposed upon return to physical activity using a randomized trial design. Women undergoing pelvic floor reconstructive surgery will be randomized to either (i) standard pre-operative education (ii) modified, patient-centered pre-operative education. The investigators will monitor both post-operative opioid consumption and return to physical activity. The investigators hypothesize that investigation of patient's post-operative pain experiences and their inclusion in the educational and the shared decision-making process will likely decrease post-operative narcotic use without affecting return to function. Our long-term goal is to develop a pragmatic and balanced approach to address pain concerns, decreasing the medical community's contribution to the opioid epidemic.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are ≥ 18 years of age
2. English or Spanish speaking
3. Patient scheduled for pelvic floor surgery

Exclusion Criteria:

1. Unable to speak English or Spanish
2. Using long acting opioids (e.g. MS Contin, Fentanyl patch)
3. Primary or Pain Healthcare Provider recommends against study participation (eg. If the patient has a history of opioid use disorder or other confounding problems, we will contact the Primary Care Provider or Pain Healthcare Provider for their recommendations regarding study participation)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuko Komesu, MD, Study Director — University of New Mexico
Locations (2):
- United States (2):
  - UNMH Women's Care Clinic, Albuquerque, New Mexico
  - UNM Sandoval Regional Medical Center, Rio Rancho, New Mexico

REFERENCES:
- [Derived] Serna-Gallegos TR, Komesu YM, Dunivan GC, Meriwether KV, Ninivaggio CS, Petersen TR, Jeppson PC. Randomized Trial on Expectations and Pain Control Advancement in Surgery: The REPAIR Study. Urogynecology (Phila). 2024 Jan 1;30(1):7-16. doi: 10.1097/SPV.0000000000001387. Epub 2023 Jun 27. PMID 37428883

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Patient Centered Pre-op Education | Routine Pre-op Education
Started | 86 | 88
Completed | 86 | 88
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Centered Pre-op Education | Routine Pre-op Education | Total
Number analyzed (Participants) | 86 | 88 | 174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 86 | 88 | 174
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 53 [40 to 65] | 55 [42 to 68] | 54 [40 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 88 | 174
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 11 | 18
  Asian | NA — It was optional for patients to give us race/ethnicity data therefore not everyone did it and the numbers do not equal the total number of participants. | NA — It was optional for patients to give us race/ethnicity data therefore not everyone did it and the numbers do not equal the total number of participants. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander | NA — It was optional for patients to give us race/ethnicity data therefore not everyone did it and the numbers do not equal the total number of participants. | NA — It was optional for patients to give us race/ethnicity data therefore not everyone did it and the numbers do not equal the total number of participants. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American | NA — It was optional for patients to give us race/ethnicity data therefore not everyone did it and the numbers do not equal the total number of participants. | NA — It was optional for patients to give us race/ethnicity data therefore not everyone did it and the numbers do not equal the total number of participants. | NA — Total not calculated because data are not available (NA) in one or more arms.
  White | 33 | 35 | 68
  More than one race | 1 | 5 | 6
  Unknown or Not Reported | 45 | 37 | 82

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use at Approximately Two Weeks Post-op
Description: Morphine milligram equivalents at the two weeks post-op
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Patient Centered Pre-op Education | Routine Pre-op Education
Number analyzed (Participants) | 86 | 88
MME | 15 [0 to 75] | 22.5 [0 to 60]

2. Secondary Outcome: Opioid Use at Approximately Six to Eight Weeks Post-op
Description: Morphine milligram equivalents at the six to eight weeks post-op
Time Frame: 6-8 weeks
Measure: Median (Inter-Quartile Range); unit: MME
Arm/Group | Patient Centered Pre-op Education | Routine Pre-op Education
Number analyzed (Participants) | 86 | 88
MME | 15 [0 to 75] | 23 [0 to 68]

ADVERSE EVENTS:
Time Frame: Enrollment of patient until 8 weeks post-operatively for each patient.
Description: All adverse events were collected routinely.
Arm/Group | Patient Centered Pre-op Education | Routine Pre-op Education
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/88
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/88
Other Adverse Events (participants affected / at risk) | 0/86 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT03726476/Prot_SAP_000.pdf